CLINICAL TRIAL: NCT01352585
Title: An Exploratory, Observational, Multicentre Study to Investigate the Impact of the Presence of JAK2 (V617F) Mutation on Treatment Response in Patients With Essential Thrombocythaemia Treated With XAGRID® (Anagrelide Hydrochloride)
Brief Title: Exploratory Multi-centre Trial In Patients With ET Treated With XAGRID®
Acronym: EMIX
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD422-703
Record Dates: First submitted 2011-05-10; First posted 2011-05-12 (Estimated); Results first posted 2014-07-29 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Essential Thrombocythemia (ET)
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — anagrelide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- JAK2 Positive Participants
  Interventions: Drug: Anagrelide hydrochloride
- JAK2 Negative Participants
  Interventions: Drug: Anagrelide hydrochloride

INTERVENTIONS:
Drug: Anagrelide hydrochloride — 0.5 mg hard capsules, dosing decisions will be made by the treating physician
  Other Names: Xagrid

SUMMARY:
This study is hypothesis-generating to explore the impact of JAK2 (V617F) mutation status on the treatment response to anagrelide hydrochloride

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be able to understand and willing to participate in the study, and provide a personally dated and signed written informed consent form.
2. Patients must have a confirmed diagnosis of ET according to the World health Organisation's criteria.
3. ET patients who are uncontrolled, in the Investigator's opinion, by first-line (or previous) cytoreductive treatment for efficacy or tolerance reasons.
4. Patients who have either commenced treatment with anagrelide hydrochloride in the last 7 days or for whom a decision has been documented to commence treatment with anagrelide hydrochloride

Exclusion Criteria:

1. Patients for whom treatment with anagrelide hydrochloride is contraindicated, according to the current XAGRID SmPC.
2. Known or suspected intolerance or hypersensitivity to the product, closely related compounds, or any of the stated ingredients.
3. Patients participating in an interventional research study.
4. Patients on combination therapy or for whom there is an intention to treat with other cytoreductive agents e.g., hydroxyurea, interferon. Patients can however use aspirin and other anti-aggregatory products at the Investigator's discretion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ET patients in Italy
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-07-19 (Actual); Primary Completion 2013-09-19 (Actual); Study Completion 2013-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (10):
- Italy (10):
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Istituto Seragnoli-Policlinico S.Orsola-Malpighi, Bologna
  - A.O. Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale San Martino, Genova
  - Fondazione IRCCS Ca' Granda, Milan
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Ospedale Maggiore della Carita, Novara
  - Policlinico A. Gemelli, Roma
  - Padiglione ex-oncologico Ospedale S.Maria, Terni

REFERENCES:
- [Result] Cascavilla N, De Stefano V, Pane F, Pancrazzi A, Iurlo A, Gobbi M, Palandri F, Specchia G, Liberati AM, D'Adda M, Gaidano G, Fjerza R, Achenbach H, Smith J, Wilde P, Vannucchi AM. Impact of JAK2(V617F) mutation status on treatment response to anagrelide in essential thrombocythemia: an observational, hypothesis-generating study. Drug Des Devel Ther. 2015 May 18;9:2687-94. doi: 10.2147/DDDT.S79576. eCollection 2015. PMID 26028965

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Started | 23 | 24
Completed | 15 | 21
Not Completed | 8 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (14.00) | 58.6 (15.94) | 58.0 (14.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 9 | 10 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Italy | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Platelet Count ≤600x10^9/L After 12 Months
Description: A platelet count of ≤600x10^9/L after 12 months is considered at least a partial response.
Time Frame: 1 year
Population: The Full Analysis Set (FAS) in each JAK2 status group who had a viable platelet sample during the 12-month follow-up window. For this Outcome Measure 35 patients in the FAS had a viable laboratory sample.
Measure: Number; unit: participants
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 14 | 21
participants | 12 | 14

2. Secondary Outcome: Number of Patients With Platelet Count ≤400x10^9/L After 12 Months
Description: A platelet count of ≤400x10^9/L after 12 months is considered a complete response.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 14 | 21
participants | 7 | 8

3. Secondary Outcome: Platelet Count
Time Frame: 1 year
Population: The Full Analysis Set (FAS) in each JAK2 status group who had a viable platelet sample during the 12-month follow-up window. For this Outcome Measure 28 patients in the FAS had a viable laboratory sample.
Measure: Mean (Standard Deviation); unit: Platelets (x10^9/L)
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 17
Platelets (x10^9/L) | 458.9 (163.25) | 503.0 (254.04)

4. Secondary Outcome: Red Blood Cell (RBC) Count
Time Frame: 1 year
Population: The Safety Analysis Set (SAS) consisted of all subjects enrolled in the study who took at least 1 dose of anagrelide hydrochloride. 27 patients in the SAS met this requirement and had a viable laboratory sample.
Measure: Mean (Standard Deviation); unit: RBC Count (x10^12/L)
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 16
RBC Count (x10^12/L) | 4.85 (0.430) | 4.24 (0.797)

5. Secondary Outcome: White Blood Cell (WBC) Count
Time Frame: 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: WBC Count (x10^9/L)
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 17
WBC Count (x10^9/L) | 7.75 (1.317) | 8.77 (3.770)

6. Secondary Outcome: Differential WBC Count - Neutrophils, Lymphocytes, Monocytes, and Basophils.
Time Frame: 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 17
percent
  Neutrophils | 62.05 (4.429) | 60.07 (13.515)
  Lymphocytes | 27.53 (4.412) | 28.76 (12.381)
  Monocytes | 6.50 (2.235) | 7.21 (2.680)
  Basophils | 1.75 (2.425) | 0.81 (0.486)

7. Secondary Outcome: Differential WBC Count - Eosinophils
Time Frame: 1 year
Population: The Full Analysis Set (FAS) in each JAK2 status group who had a viable platelet sample during the 12-month follow-up window. For this Outcome Measure 27 patients in the FAS had a viable laboratory sample.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 16
percent | 2.95 (1.958) | 2.77 (1.906)

8. Secondary Outcome: Hemoglobin Concentration
Time Frame: 1 year
Population: The Safety Analysis Set (SAS) consisted of all subjects enrolled in the study who took at least 1 dose of anagrelide hydrochloride. 28 patients in the SAS had a viable laboratory sample.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 17
g/L | 133.6 (13.09) | 120.2 (16.85)

9. Secondary Outcome: Hematocrit Level
Description: The proportion of the volume of red blood cells to the total volume of blood.
Time Frame: 1 year
Population: The Safety Analysis Set (SAS) consisted of all subjects enrolled in the study who took at least 1 dose of anagrelide hydrochloride. 27 patients in the SAS had a viable laboratory sample.
Measure: Mean (Standard Deviation); unit: Hematocrit (fraction of 1)
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Number analyzed (Participants) | 11 | 16
Hematocrit (fraction of 1) | 0.412 (0.0335) | 0.367 (0.0608)

ADVERSE EVENTS:
Arm/Group | JAK2 Positive Participants | JAK2 Negative Participants
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 6/23 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JAK2 Positive Participants (N=23) | JAK2 Negative Participants (N=24)
anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Scotoma (Eye disorders) | 0 | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 4 (4)
Presyncope (Nervous system disorders) | 1 (1) | 0
Dermatits (Skin and subcutaneous tissue disorders) | 1 (1) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.